CLINICAL TRIAL: NCT01310335
Title: Effect of Whole-Body Vibration on Plasma Sclerostin Level in Healthy Young Adult Women
Brief Title: Effect of Whole-Body Vibration on Plasma Sclerostin Level
Acronym: WBV-SCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan Karacan, Clinical Associated Professor, Chief of Physical Med & Rehab Clinic, Bagcilar Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BEAH FTR-1
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Osteopenia
Keywords: sclerostin; whole-body vibration
MeSH Terms: conditions — Bone Diseases, Metabolic; Sclerosteosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Training (Experimental): The whole-body vibration (WBV) training
  Interventions: Device: whole-body vibration (WBV)

INTERVENTIONS:
Device: whole-body vibration (WBV) — All cases will be trained on a whole-body vibration (WBV) platform (Power Plate) 5 times a week for one week period.
  Other Names: Cyclic mechanical loading

SUMMARY:
The aim of this study is to investigate effect of whole-body vibration on plasma sclerostin level in healthy young adult women.

Fifteen healthy young adult women are planned to include in this study. All cases will be trained on a whole-body vibration (WBV) platform (Power Plate) 5 times a week for one week period. Training duration will be short at the beginning but progressed slowly.

The amplitude of vibration will be 2 mm and the frequency of the vibration will be 40 Hz. The subjects will be asked to report negative side effects or adverse reactions in their training diary.

Previbration and postvibration (just after, 10.minute and 30.minute) levels of plasma sclerostin will be measured on first, second and fifth day of experiment. Sclerostin levels will be measured by human sclerostin ELISA kit.

DETAILED DESCRIPTION:
Whole-body vibration has a strong osteogenic effect. The cyclic mechanical loading to the bone stimulates the osteocytes.

Sclerostin, the protein product of the SOST gene, is an osteocyte-specific cysteine knot-secreted glycoprotein that is a potent inhibitor of bone formation. Sost/sclerostin levels have been reported to be reduced by mechanical stimulation.

The aim of this study is to investigate effect of whole-body vibration on plasma sclerostin level in healthy young adult women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women,
* Women with ages varying between 20 and 40 years
* Right-handed women

Exclusion Criteria:

* Lower extremity problems

  1. Orthopedic problems: shortness of legs, congenital anomalies, etc.
  2. Joint disease (arthritis, joint prosthesis, etc.)
  3. Other painful pathologies in the lower extremities (fractures, tendinitis,bursitis, etc.)
  4. Circulation problems in the lower extremities
* Dorsolumbar diseases: Vertebral fract, disc hernias, spondylodiskitis, etc.
* Systemic disease cases

  1. Systemic bone disease: osteoporosis, osteomalacia, Paget's disease
  2. Hypertension (>135 mmHg systolic, >85 mmHg diastolic)
  3. Heart dis.(coronary dis, conduction/rhythm prob, cardiac pacemaker)
  4. Infectious diseases
  5. Endocrine diseases (Diabetes mellitus etc)
* Neurological diseases (CNS problems, peripheral neuropathy)
* Menstrual cycle disorders, amenorrhea, lactation, oral contraceptive use
* Cases during the ovulatory period (11-16th day of menses)
* Obesity (BMI >30 kg/m2) or low BMI (BMI <20 kg/m2)
* Vertigo
* Cognitive function disorders
* Women whose blood samples were not taken in the time planned
* Women whose blood samples hemolyzed

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Plasma Sclerostin Level | 1 month
  Change of plasma sclerostin level with whole-body vibration

CONTACTS AND LOCATIONS:
Overall Officials: ILHAN KARACAN, MD, Study Chair — Bagcilar Training & Research Hospital
Locations (1):
- Bagcilar Training & Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No